CLINICAL TRIAL: NCT01527253
Title: Effects of a Synergistic Food Basket on Markers of Metabolic Syndrome Risk in Healthy Mature Women
Brief Title: Effect of a Synergistic Food Basket on Metabolic Syndrome Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Juscelino Tovar, Project Manager, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AFC-Food Basket
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Metabolic Syndrome; Insulin Resistance
Keywords: Cardiometabolic risk; Metabolic syndrome; Prebiotics; Legumes; Wholegrain cereal; Functional diet; Low glycemic index diet
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Diet (Experimental): Subjects eat a diet designed according to the Nordic Dietary Recommendations containing important amounts of specific legume and cereal ingredients that provide substrates for the intestinal microflora (prebiotics)
  Interventions: Other: Synergistic food basket
- Control diet (Experimental): Subjects eat a diet designed according to the Nordic Dietary Recommendations but lacks the specific legume and cereal ingredients that provide substrates for the intestinal microflora (prebiotics).
  Interventions: Other: Synergistic food basket

INTERVENTIONS:
Other: Synergistic food basket — A low glycemic index diet enriched in dried legumes and wholegrain cereals is compared with a control regime lacking these functional ingredients for their ability to ameliorate different markers associated with the risk for developing cardiometabolic disease

SUMMARY:
The study evaluates the effect of a diet combining two different functional concepts on markers associated to cardiometabolic risk. The functional concepts are selected on the basis of their reported ability to influence the inflammatory tonus. It is hypothesized that the medium-term consumption of a diet combining low GI-prebiotic foods may positively influence various biomarkers associated with the risk for developing metabolic syndrome and cardiometabolic disease. Also, the combination of functional mechanisms are expected to result in synergistic effects.

DETAILED DESCRIPTION:
The intervention is carried out in healthy women following a randomized crossover design in which an "active" (functional") diet is compared with a control diet formulated in agreement with the Nordic Dietary Recommendations but lacking the functional ingredients of the active regime.

The active diet supplies important daily amounts of dried legumes and wholegrain cereal products.

Each dietary treatment is applied for 4 weeks separated by a 4-6 week washout period. Subjects are encouraged to maintain a stable body weight under the whole trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 32 kg/m2

Exclusion Criteria:

* Fasting blood glucose > 6.1 mmol/L
* Medication for high blood pressure and/or elevated blood cholesterol

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LDL cholesterol after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)

SECONDARY OUTCOMES:
Change from baseline in LDL-cholesterol/HDL-cholesterol after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in fasting plasma triglycerides after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in fasting CRP after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in fasting plasma PYY after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
  Satiety signalling hormone PYY
Change from baseline in fasting plasma insulin after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in fasting plasma glucose after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in fasting plasma PAI-1 after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in BMI after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
  Body Mass Index
Change from baseline in blood pressure after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in HOMA-IR after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)
Change from baseline in waist circumference after each dietary period | Week 0 and after 4 weeks (Start and End of the intervention arm)

CONTACTS AND LOCATIONS:
Overall Officials: Inger Björck, PhD Prof., Study Chair — Antidiabetic Food Centre, Lund University; Juscelino Tovar, PhD, Study Director — Antidiabetic Food Centre, Lund University; Anne Nilsson, PhD, Principal Investigator — Lund University; Maria Johansson, PhD, Principal Investigator — Antidiabetic Food Centre, Lund University
Locations (1):
- Antidiabetic Food Centre, Chemical Centre. Lund University, Lund, Skåne County, Sweden

REFERENCES:
- [Background] Nilsson A, Ostman E, Preston T, Bjorck I. Effects of GI vs content of cereal fibre of the evening meal on glucose tolerance at a subsequent standardized breakfast. Eur J Clin Nutr. 2008 Jun;62(6):712-20. doi: 10.1038/sj.ejcn.1602784. Epub 2007 May 23. PMID 17522615
- [Background] Nilsson AC, Ostman EM, Holst JJ, Bjorck IM. Including indigestible carbohydrates in the evening meal of healthy subjects improves glucose tolerance, lowers inflammatory markers, and increases satiety after a subsequent standardized breakfast. J Nutr. 2008 Apr;138(4):732-9. doi: 10.1093/jn/138.4.732. PMID 18356328
- [Background] Nilsson AC, Ostman EM, Granfeldt Y, Bjorck IM. Effect of cereal test breakfasts differing in glycemic index and content of indigestible carbohydrates on daylong glucose tolerance in healthy subjects. Am J Clin Nutr. 2008 Mar;87(3):645-54. doi: 10.1093/ajcn/87.3.645. PMID 18326603
- [Background] Liljeberg HG, Akerberg AK, Bjorck IM. Effect of the glycemic index and content of indigestible carbohydrates of cereal-based breakfast meals on glucose tolerance at lunch in healthy subjects. Am J Clin Nutr. 1999 Apr;69(4):647-55. doi: 10.1093/ajcn/69.4.647. PMID 10197565
- [Result] Tovar J, Nilsson A, Johansson M, Bjorck I. Combining functional features of whole-grain barley and legumes for dietary reduction of cardiometabolic risk: a randomised cross-over intervention in mature women. Br J Nutr. 2014 Feb;111(4):706-14. doi: 10.1017/S000711451300305X. Epub 2013 Sep 24. PMID 24063257